CLINICAL TRIAL: NCT06313424
Title: Arthroscopic Treatment of Meniscal Lesions on Healthy Meniscus in Children and Adolescents: Diagnostic Circumstances, Treatment and Results
Brief Title: Arthroscopic Treatment of Meniscal Lesions on Healthy Meniscus in Children and Adolescents
Acronym: ATML
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9029
Record Dates: First submitted 2024-01-05; First posted 2024-03-15 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-01

CONDITIONS: Knee Injuries
Keywords: Knee Injuries; Meniscus; Pediatric traumatology
MeSH Terms: conditions — Knee Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Meniscal lesions are common in pediatrics and mainly affect adolescents. These lesions can jeopardize the functional prognosis of the knee in the short, medium or long term if they are not well managed.

More precisely, it is a question of determining whether arthroscopic repair of isolated meniscal lesions in children gives good results and what factors influence them, with the aim of improving the care of children suffering from meniscal lesions.

The treatment of meniscal lesions comes down to either conservative or restorative treatment or non-conservative treatment by meniscectomy. For most authors, the treatment of meniscal lesions must remain restorative through meniscal suture, leaving no room for meniscectomy. The open approach has given way to the arthroscopic approach which, according to the literature, is the gold standard. Meniscal lesions are varied and therefore there are numerous therapeutic procedures. Therapeutic indications are precise but the results of the treatments remain differently assessed depending on the studies; studies evaluating the results of treatment in the pediatric population are few in number.

Based on this observation, the present study aims to describe the results of repairs of meniscal lesions in pediatric traumatology.

ELIGIBILITY:
Inclusion Criteria:

* Minor subject under 18 years old
* Subject operated on at Strasbourg University Hospital for repair of lesions on healthy meniscus during the period from February 1, 2010 to September 30, 2022.
* Absence of written opposition in the medical file of the subject (and/or their legal representative if applicable) to the reuse of their data for scientific research purposes.

Exclusion Criteria:

* Presence of opposition from the subject (and/or their legal representative if applicable) to the reuse of their data for scientific research purposes.
* Subject with lesion on discoid meniscus
* Incomplete or unusable clinical file

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Minor subject (under 18 years old) operated on at Strasbourg University Hospital for repair of lesions on healthy meniscus during the period from February 1, 2010 to September 30, 2022.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-08-29 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-04-29 (Estimated)

PRIMARY OUTCOMES:
description of the results of repairs of meniscal lesions in pediatric traumatology | Files analysed retrospectively from February 1, 2010 to September 30, 2022 will be examined
  This study is retrospective

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Chirurgie Pédiatrique - CHU de Strasbourg - France, Strasbourg, France